CLINICAL TRIAL: NCT05462197
Title: The Influence of Qigong Wuqinxi on Chronic Pain, Sleep Quality, Traditional Chinese Medical Body Constitution, and Tongue Features of the Community-Dwelling Older Adults
Brief Title: The Influence of Qigong Wuqinxi on Health Status of the Community-Dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Tzu-wei Chou, research project leader, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-049-B
Record Dates: First submitted 2022-07-02; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Sleep Quality; Chronic Pain
Keywords: Qigong Wuqinxi; Chronic Pain; Sleep Quality; Traditional Chinese Medical Body Constitution; Tongue Features; Community-Dwelling Older Adults
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong Wuqinxi group (Experimental): The Wuqinxi version adopted by this research is the Health Qigong Wuqinxi newly compiled in mainland China in 2003. There are only 10 movements in total. It is practiced three times a week for 3 months, including group practice once a week, 50 minutes each time, and the other two times of independent practice, the same 50 minutes each time, and the practice form must be filled out.
  Interventions: Behavioral: Qigong Wuqinxi
- control group (No Intervention): The control group was carried out according to the original daily activities without any intervention activities

INTERVENTIONS:
Behavioral: Qigong Wuqinxi — Wuqinxi is an exercise method developed by the ancient Chinese physician Hua Tuo by combining the ancient guide, breathing, and imitating the shapes of five animals, such as tiger, deer, bear, ape, and bird, combined with the zang-fu and meridian theory of traditional Chinese medicine. There have been studies in the past proven that this exercise can achieve health-promoting effects
  Arms: Qigong Wuqinxi group

SUMMARY:
Pain and sleep disturbance are common symptoms of community-dwelling older adults observed in traditional Chinese medical(TCM) clinics. Acupuncture or other medical treatments have their side effects and usage limitations, so it is expected that other non-medical interventions can relieve the symptoms. The purpose of this study was to test the effect of Qigong Wuqinxi intervention on pain, sleep quality, TCM body constitution and tongue features of the community-dwelling older adults.

DETAILED DESCRIPTION:
Methods: using cluster randomised clinical trial , two community care sites in Sanmin District, Kaohsiung City were selected. Community-dwelling older adults who are over 65 years old and have the ability to communicate in Mandarin and Taiwanese were recruited . Those who had severe mental illness, moderate to severe dementia (level 2 or above on the Clinical Dementia Assessment Scale) and Barthel Index score <60 were excluded. There were 63 valid cases divided into experimental group(n=32) and control group(n=31). The experimental group practiced Qigong Wuqinxi 50 minutes three times a week for 12 weeks; meanwhile, the control group maintained routine daily activities. The two groups of participants were tested before and after the intervention period with the following research tools: 1) The Brief Pain Inventory, (BPI), 2) Pittsburgh Sleep Quality Index (PSQI), 3) Body Constitution Questionnaire (BCQ), 4) automatic tongue diagnosis system (ATDS). The research data were analyzed with SPSS 19 software package for descriptive statistics, chi-square test, independent t test and paired t test.

ELIGIBILITY:
Inclusion Criteria:

* 65-85 year olds
* have the ability to communicate in Mandarin and Taiwanese and can answer questions orally

Exclusion Criteria:

* severe mental illness,
* moderate to severe dementia (Clinical Dementia Assessment Scale Level 2 or above)
* almost unable to perform daily activity by self. (Barthes scale <60)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
musculoskeletal chronic pain | 1 month
  musculoskeletal chronic pain of the Community-Dwelling Older Adults assessed byThe Brief Pain Inventory (BPI) [ Developed by Cleeland (1985). The pain scale has a clear human-shaped image, a total of 20 items, and the content is divided into pain intensity and pain interference subscales. The scale uses a scale of 0-10, with a pain score of 0 being no pain, 1-4 being mild pain, 5-6 being moderate pain, and 7-10 being severe pain. Good reference indicator. This scale has been widely used and translated into more than ten languages and has good reliability and validity. Ger et al. (1999) translated this scale into the Brief Pain Inventory-Taiwanese Version (BPI-T) ]
health status | 1 month
  health status of the Community-Dwelling Older Adults assessed by Body Constitution Questionnaire,BCQ.[The "Traditional Chinese medicine constitution type and constitution scoring rule table" is used to analyze the patient's constitution type, and classify and classify according to the constitution scoring rules. The five-point Likert scale was used for each question, and words suitable for the frequency and intensity of the case were selected. BCQ Constitution Questionnaire: A total of 44 questions, including: 19 questions for Yin deficiency, the standard for yin deficiency constitution is more than 30 points; 19 questions for Yang deficiency, the scoring standard is more than 31 points; 16 questions for phlegm-dampness and blood stasis constitution, the judgment standard The standard is more than 27 points. If the total score does not meet the criteria for any of the three constitutions, it does not belong to any of the three constitutions, and is defined as "peaceful constitution".
Tongue Features | 1 month
  Tongue Features of the Community-Dwelling Older Adults assessed by Automatic Tongue Diagnosis System (ATDS) . [ ATDS can identify nine main features, namely tongue color, tongue coating color, tongue coating thickness (ratio of thick coating), body fluid, tongue shape, cracks, vermilion spots, ecchymoses and tooth marks, to generate information about length (cm), area ( cm²), humidity and details of the number of cracks, dents, red dots. ATDS can capture tongue images and automatically and reliably extract features to assist TCM practitioners in diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Chen k Min, Professor, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Master Program of Long-Term Care in Aging of Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo Y, Xu M, Wei Z, Hu Q, Chen Y, Yan J, Wei Y. Beneficial Effects of Qigong Wuqinxi in the Improvement of Health Condition, Prevention, and Treatment of Chronic Diseases: Evidence from a Systematic Review. Evid Based Complement Alternat Med. 2018 Oct 24;2018:3235950. doi: 10.1155/2018/3235950. eCollection 2018. PMID 30473716
- [Background] Wei X, Xu A, Yin Y, Zhang R. The potential effect of Wuqinxi exercise for primary osteoporosis: A systematic review and meta-analysis. Maturitas. 2015 Dec;82(4):346-54. doi: 10.1016/j.maturitas.2015.08.013. Epub 2015 Sep 19. PMID 26386831
- [Derived] Chou TW, Kuo CC, Chen KM, Belcastro F. Influence of Qigong Wuqinxi on Pain, Sleep, and Tongue Features in Older Adults. J Nurs Res. 2024 Dec 1;32(6):e358. doi: 10.1097/jnr.0000000000000646. PMID 39593225